CLINICAL TRIAL: NCT02391623
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Multiple Escalating Oral Doses Of Pf-06427878 Co Administered With And Without Food In Healthy Adult Subjects
Brief Title: A Multiple Oral Doses Study Of PF-06427878 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7871002; 2015-000130-29 (EudraCT Number)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Subjects
Keywords: Multiple Ascending Dose; Healthy Subjects; Hyperlipidemia; Lipid Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Hyperlipidemias; Lipid Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Single dose level of PF-06427878 at 5 mg or placebo every 8 hours (Q8H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06427878; Drug: Placebo
- Cohort 2 (Experimental): Single dose level of PF-06427878 at a dose no more than 3.5-fold increase from Cohort 1 or placebo every 8 hours (Q8H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06427878; Drug: Placebo
- Cohort 3 (Experimental): Single dose level of PF-06427878 at a dose no more than 3.5-fold increase from Cohort 2 or placebo every 8 hours (Q8H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06427878; Drug: Placebo
- Cohort 4 (Experimental): Single dose level of PF-06427878 at a dose no more than 3.5-fold increase from Cohort 3 or placebo every 8 hours (Q8H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06427878; Drug: Placebo
- Cohort 5 (Experimental): Single dose level of PF-06427878 at a dose no more than 3.5-fold increase from Cohort 4 or placebo every 8 hours (Q8H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06427878; Drug: Placebo
- Cohort 6 (Experimental): Single dose level of PF-06427878 (with the same total daily dose as Cohort 5) or placebo every 12 hours (Q12H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06427878; Drug: Placebo

INTERVENTIONS:
Drug: PF-06427878 — PF-06427878 will be administered as an extemporaneously prepared solution every 8 hours for 14 days (n=8).
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5
Drug: Placebo — Placebo will be administered as an extemporaneously prepared solution every 8 hours for 14 days (n=2).
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5
Drug: PF-06427878 — PF-06427878 will be administered as an extemporaneously prepared solution every 12 hours for 14 days (n=8).
  Arms: Cohort 6
Drug: Placebo — Placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days (n=2).
  Arms: Cohort 6

SUMMARY:
PF-06427878 is a new compound proposed for the treatment of hyperlipidemia. The primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of multiple oral doses of PF-06427878 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential.
* Body Mass Index (BMI) of 17.5 to 35.4 kg/m2; and a total body weight >50 kg
* Subjects with fasting TG level of >=90 mg/dL and <=500 mg/dL following an overnight fast
* Subjects with low density lipoprotein cholesterol between 115 mg/dL and 190 mg/dL following an overnight fast

Exclusion Criteria:

•Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs). | 0-25 days
Assessment of clinical laboratory tests. | 0-25 days
Assessment of vital signs (including blood pressure and pulse rate). | 0-25 days
Assessment of cardiac conduction intervals as assessed via 12-lead electrocardiogram (ECG). | 0-25 days

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 1 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06427878during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 12 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06427878 on day 14 | 0, 1, 2, 3, 4, 6, 8, 12 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 1 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 12 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Area Under the Curve for PF-06427878 during the dosing interval (AUCtau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 1 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Area Under the Curve for PF-06427878 during the dosing interval (AUCtau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 12 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Area Under the Curve for PF-06427878 during the dosing interval (AUCtau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Plasma Decay Half-Life (t1/2) for PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Apparent Volume of Distribution (Vz/F) of PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Apparent Oral Clearance (CL/F) of PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Minimum Observed Plasma Concentration (Cmin) for PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Peak:Trough ratio of PF-06427878 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Accumulation ratio for Maximum Observed Plasma Concentration (Rac(Cmax)) for PF-06427878 on day14 relative to day 1 | 0, 1, 2, 3, 4, 6, 8, 12 hours post dose
Accumulation ratio for Maximum Observed Plasma Concentration (Rac(Cmax)) for PF-06427878 on day14 relative to day 1 during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Accumulation ratio for Area Under the Curve during the dosing interval (Rac(AUCtau)) for PF-06427878 on day14 relative to day 1 | 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post dose
Amount of PF-06427878 excreted in urine (Ae) during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0- tau hours post dose
Percent of dose excreted in urine as PF-06427878 (Ae%) during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0- tau hours post dose
Renal clearance of PF-06427878 (CLr) during the dosing interval (tau), ie, 0-8H for Q8H, 0-12H for Q12H, and 0-24H for QD, on day 14 | 0- tau hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Amin NB, Carvajal-Gonzalez S, Purkal J, Zhu T, Crowley C, Perez S, Chidsey K, Kim AM, Goodwin B. Targeting diacylglycerol acyltransferase 2 for the treatment of nonalcoholic steatohepatitis. Sci Transl Med. 2019 Nov 27;11(520):eaav9701. doi: 10.1126/scitranslmed.aav9701. PMID 31776293
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7871002&StudyName=A%20Phase%201%2C%20Randomized%2C%20Double-blind%2C%20Placebo-controlled%20Study%20To%20Assess%20The%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetics%20Of%20Multiple%20Escalating%20Oral%20Doses%20Of%20Pf-06427878%20Co%20Administered%20With%20And%20Without%20Food%20In%20Healthy%20Adult%20Subjects